CLINICAL TRIAL: NCT04672824
Title: A Phase I Study to Determine the Safety and Immunogenicity of the Candidate Rift Valley Fever Virus (RVFV) Vaccine ChAdOx1 RVF Among Healthy Adult Volunteers in Uganda
Brief Title: A Study to Assess the New Candidate Rift Valley Fever Virus Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: RVF002
Record Dates: First submitted 2020-10-19; First posted 2020-12-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-01

CONDITIONS: RVF; Rift Valley Fever
Keywords: Rift Valley Fever; Vaccine; ChAdOx1
MeSH Terms: conditions — Rift Valley Fever | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ChAdOx1 RVF group 1 (Experimental): Participants will receive ChAdOx1 RVF 5 x 10^9 vp, delivered intramuscularly
  Interventions: Biological: ChAdOx1 RVF
- Control group (Active Comparator): Placebo (Normal Saline), 0.5ml delivered intramuscularly
  Interventions: Other: Saline
- ChAdOx1 RVF group 2 (Experimental): Participants will receive ChAdOx1 RVF 2.5 x 10^10 vp, delivered intramuscularly
  Interventions: Biological: ChAdOx1 RVF
- ChAdOx1 RVF group 3 (Experimental): Participants will receive ChAdOx1 RVF 5 x 10^10 vp, delivered intramuscularly
  Interventions: Biological: ChAdOx1 RVF

INTERVENTIONS:
Biological: ChAdOx1 RVF — Single dose ChAdOx1 vectored vaccine
  Arms: ChAdOx1 RVF group 1; ChAdOx1 RVF group 2; ChAdOx1 RVF group 3
Other: Saline — 0.5ml saline placebo
  Arms: Control group

SUMMARY:
Randomised, single blind, placebo - controlled, dose-escalation, phase I clinical trial recruiting healthy adults aged 18-50 years

DETAILED DESCRIPTION:
This is a randomised, single blind, placebo-controlled, dose escalation, phase I clinical trial to assess the safety and immunogenicity of the candidate ChAdOx1 RVF vaccine in healthy Ugandan volunteers aged 18-50. The vaccine will be administered intramuscularly.

This study will run concurrently with the first-in-human ChAdOx1 RVF trial in Oxford. Vaccination at the MRC/UVRI and LSHTM Uganda Research Unit, Masaka will only begin upon receiving a favourable opinion of Uganda's trial DSMB of the 7-day post-vaccination safety analysis of the first two lowest dose groups (ChAdOx1 RVF 5 x 10^9vp and ChAdOx1 RVF 2.5 x 10^10vp) of the trial in Oxford.

Volunteers will be recruited and vaccinated at the MRC/UVRI and LSHTM Uganda Research Unit Clinical Research Centre in Masaka. There will be three study groups and a total of 30 volunteers will be enrolled (table 3). Volunteers will be recruited sequentially into Groups 1,2 and 3. Within each group, eligible volunteers will be randomly allocated to receive either ChAdOx1 RVF or placebo of 0.9% Normal Saline in a ratio of 2:1 in group 1 and 5:1 in groups 2 and 3. The DSMB will analyse the 7-day post-vaccination safety data in each group and advise on whether to proceed to the next group with a higher dose .

ELIGIBILITY:
Inclusion Criteria:

The volunteer must satisfy all the following criteria to be eligible for the study:

1. Male and female healthy adults aged 18 to 50 years
2. Able and willing to provide written informed consent
3. Able and willing (in the Investigator's opinion) to comply with all study requirements
4. For females only, willingness to practice continuous effective contraception during the study.
5. Females of childbearing potential must have a negative urine β-human chorionic gonadotropin (β-hCG) pregnancy test at screening and a negative urine β-hCG pregnancy test immediately prior to study vaccine administration
6. Agreement to refrain from blood donation during the course of the study
7. Healthy in the investigator's clinical judgement basing on the medical history and physical examination performed at screening
8. Healthy on the basis of clinical laboratory tests (within the institutional normal laboratory reference ranges) performed at screening.
9. Willing to provide verifiable identification to the study team
10. Volunteer must have a means to be contacted or be willing to provide locator information to the study team
11. Volunteer must pass the Test of Understanding (TOU)

Exclusion Criteria:

The volunteer may not enter the study if any of the following apply:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational vaccine as it may impact on interpretation of the trial data.
3. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
4. Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed)
5. History of allergic disease or reactions likely to be exacerbated by any component of the vaccine
6. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
7. Any history of anaphylaxis in relation to vaccination
8. Pregnancy, lactation or willingness/intention to become pregnant during the study
9. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
10. History of serious psychiatric condition likely to affect participation in the study
11. Bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venepuncture
12. Acute illness or temperature ≥37.5°C/99.5°F on the day of vaccination. Volunteer may be rescheduled for enrolment at a later date.
13. Major surgery (per the investigator's judgement) within 4 weeks prior to screening or planned major surgery through the course of the study
14. Any other serious chronic illness requiring hospital specialist supervision
15. Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 14 units every week
16. Suspected or known injecting drug abuse in the 5 years preceding enrolment
17. Seropositive for hepatitis B surface antigen (HBsAg)
18. Seropositive for hepatitis C virus (antibodies to HCV)
19. Any clinically significant abnormal finding on screening biochemistry, haematology and coagulation blood tests or urinalysis
20. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data
21. Prior natural exposure to RVFV as determined by seropositivity for RVFV antigens by ELISA.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile of the candidate vaccine ChAdOx1 RVF in healthy adult volunteers in Uganda: AE | The study duration: 3 months from vaccination
  Occurrence of solicited local reactogenicity signs and symptoms for 7 days following the vaccination, occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination, occurrence of unsolicited adverse events for 28 days following the vaccination, and occurrence of serious adverse events during the whole study duration
Assess the safety profile of the candidate vaccine ChAdOx1 RVF in healthy adult volunteers in Uganda: change in baseline: AE | The study duration: 3 months from vaccination
  Change from baseline for safety laboratory measures: clinical blood test adverse events (full blood count, liver function tests and renal function) graded on a scaled adapted from the FDA healthy volunteer vaccine scale

SECONDARY OUTCOMES:
Assess the immunogenicity of the candidate vaccine ChAdOx1 RVF in healthy adult volunteers in Uganda: GnGc protein antibodies | The study duration: 3 months from vaccination
  Measures of immunogenicity to the ChAdOx1 RVF vaccine:
  * ELISA to quantify antibodies to GnGc proteins
Assess the immunogenicity of the candidate vaccine ChAdOx1 RVF in healthy adult volunteers in Uganda: RVFV neutralising antibodies | The study duration: 3 months from vaccination
  Measures of immunogenicity to the ChAdOx1 RVF vaccine:
  * RVFV neutralising antibody titres
Assess the immunogenicity of the candidate vaccine ChAdOx1 RVF in healthy adult volunteers in Uganda: ELISpot & flow cytometry | The study duration: 3 months from vaccination
  Measures of immunogenicity to the ChAdOx1 RVF vaccine:
  * Ex vivo ELISpot and flow cytometry responses to GnGc

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, PhD, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (1):
- MRC/UVRI and LSHTM Uganda Research Unit, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anywaine Z, Serwanga J, Ggayi AM, Abaasa AM, Wright D, Gombe B, Ejou P, Namata T, Kigozi A, Tukamwesiga N, Basajja V, Ankunda V, Mulondo DJ, Nambaziira F, Kakande A, Kakeeto W, Nabaggala P, Jenkin D, Lawrie A, Folegatti P, Tran N, Hansen C, Elliott AM, Hill AVS, Warimwe GM, Kaleebu P. Safety, tolerability, and immunogenicity of the ChAdOx1 RVF vaccine against Rift Valley fever among healthy adults in Uganda: a single-centre, single-blind, randomised, placebo-controlled, dose-escalation, phase 1 trial. Lancet Infect Dis. 2025 Nov 11:S1473-3099(25)00565-1. doi: 10.1016/S1473-3099(25)00565-1. Online ahead of print. PMID 41237791